CLINICAL TRIAL: NCT00203060
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group, Phase III Clinical Trial For The Efficacy, Tolerability And Safety Of Two Doses Of Rasagiline Mesylate In Early Parkinson's Disease (PD) Patients Not Treated With Levodopa
Brief Title: Effectiveness, Tolerability and Safety of Rasagiline in Early Parkinson's Disease Patients Not Treated With Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: J. Michael Nicholas, Ph.D. Sr. Director, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TVP-1012/232
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Rasagiline treatment
  Interventions: Drug: Rasagiline Mesylate
- B (Placebo Comparator): placebo arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rasagiline Mesylate — tablet, 1 or 2 mg, daily, 58 weeks
  Arms: A
Drug: placebo — tablet, once daily, 58 weeks
  Arms: B

SUMMARY:
Study to look at the effectiveness, tolerability and safety of two doses of Study Medication in Early Parkinson's Disease (PD) Patients who have not been treated with Levodopa.

ELIGIBILITY:
Inclusion Criteria:

Men and women with Parkinson's disease (PD) whose diagnosis is confirmed by at least two of the cardinal signs (resting tremor, bradykinesia, rigidity) being present, without other known or suspected cause of parkinsonism.

Subjects must be age 35 years or older.

Subjects not taking or requiring anti-parkinsonian medications, except for anticholinergics.

Exclusion Criteria:

Subjects with unstable systemic medical problems or clinically significant malignancy, with particular attention to clinically significant or unstable vascular disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 1997-07; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the safety and efficacy of rasagiline in PD subjects, not receiving or requiring carbidopa/levodopa therapy. The primary efficacy measure will be the change in total UPDRS score, calculated from baseline to 26 weeks. | 58 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Oren, MD, Study Director — Teva Pharmaceutical Industries, Ltd.